CLINICAL TRIAL: NCT02411734
Title: Effect of Executive Dysfunction on Rehabilitation Potential
Acronym: Executive
Status: Terminated | Type: Observational
Why Stopped: Administrative problems with study director
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Pro 00018268
Record Dates: First submitted 2014-12-11; First posted 2015-04-08 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Peer Review, Research
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Rehabilitation — Rehabilitation after hospitalization

SUMMARY:
Executive function will be tested in patients admitted for rehabilitation and correlated with rehabilitation success

DETAILED DESCRIPTION:
1. Rationale: Many patients who were hospitalized benefit from rehabilitation after they are discharged. Rehabilitation may be provided in one of several settings, including home, nursing home or facility specializing in rehabilitation. Success of rehabilitation depends on patient's ability and willingness to cooperate with rehabilitation staff. Unfortunately, some patients cannot or do not follow the rehabilitation protocol. If they do not participate in rehabilitation for at least 90 minutes/day, they have to be discharged from a rehabilitation facility. It would be useful to be able to predict which patients will have problem with rehabilitation after they are admitted from an acute care setting. In this study, the investigators will test the hypothesis that executive function is important for achieving rehabilitation goals.
2. Background: Executive function is a set of mental processes that helps connect past experience with present action. People use it to perform activities such as planning, organizing, strategizing, paying attention to and remembering details, and managing time and space. Executive function was the most important factor for level of care elderly individuals required (Royall, Chiodo, & Polk, 2005). This study also found that many elderly individuals have impaired executive function even though they have normal cognitive function. Executive function is also related to functional abilities in individuals with mild dementia (Martyr & Clare, 2012).
3. The research question: The hypothesis tested in this study is that rehabilitation potential is decreased in persons with impaired executive function. The purpose of this study is to attempt development of a screening tool that could be used before the patients are admitted for rehabilitation. Results of this screening would alert the rehabilitation facility about possible problems occurring after the patient is admitted for rehabilitation. If such a testing will show that patient's executive function is impaired, rehabilitation results may be improved by treatment of this impairment (Royall et al., 2009).
4. Study design: During admission of a patient, Dennise Fernandez will ask patients to state why they need rehabilitation. If they are able to state the reason, Dennise Fernandez will explained the study to them and if the patient is interested she will give him/her the Informed Consent Form. If the patient will be unable to state the reason for rehabilitation, the study will be explained to his/her proxy and informed consent given to the proxy. The patient/proxy will have time to read the Informed Consent on his/her own and ask any questions he/she may have. It the patient/proxy signs the Informed Consent, Dennise Fernandez will ask how old the patient is and the patient will be asked to complete the Trail Making Tests.

   Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). The patient should be instructed to connect the circles as quickly as possible, without lifting the pen or pencil from the paper. Time the patient as he or she connects the "trail." If the patient makes an error, point it out immediately and allow the patient to correct it. Errors affect the patient's score only in that the correction of errors is included in the completion time for the task. It is unnecessary to continue the test if the patient has not completed both parts after five minutes have elapsed.

   Step 1: Give the patient a copy of the Trail Making Test Part A worksheet and a pen or pencil. Step 2: Demonstrate the test to the patient using the sample sheet (Trail Making Part A - SAMPLE). Step 3: Time the patient as he or she follows the "trail" made by the numbers on the test.

   Step 4: Record the time. Step 5: Repeat the procedure for Trail Making Test Part B.

   Scoring:

   Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment. The patient will participate in therapy during their stay, with their participation evaluated by a) amount of time participating in therapy each day, b) need for encouragement by staff to participate. Encouragement will be rated on four point scale: i) no encouragement, ii) minimal encouragement, iii) moderate encouragement, iv) maximum encouragement. 72 hours prior to discharge, they will be asked by Dennise Fernandez to complete again Trail Making Tests.
5. Sample size: 100 patients
6. Study population: All admitted patients who will meet inclusion criteria will be approached until 100 of them signs the Informed Consent Form.

   Inclusion criteria:
   1. Admitted for rehabilitation
   2. 65 years old or older
   3. Speaks English

   Exclusion criteria:
   1. Unable to read (even with glasses)
   2. Unable to write
7. The expected results of the research: Results of this study will be published in a scientific journal. If the results are positive, a scale will be developed that will inform rehabilitation facility about rehabilitation potential of a patient before he/she is admitted for rehabilitation.
8. Principal Investigator: Ladislav Volicer, MD, PhD
9. Potential risk to the subjects: The research will not influence rehabilitation of the patients. The only risk is that they may become frustrated if they difficulty accomplishing the Trail Making Tests.
10. Experimental Procedures: Administration of the Trail Making Tests and recording duration of rehabilitation and possible need for encouragement. Results of Trail Making Test with be correlated with level of participation in therapy.
11. Potential benefit to subjects: None
12. Human subjects considerations: Informed consent will be given to patients only after they express interest in research and they will have one day to decide if they want to sign it. If a patient cannot explain the reason for his/rehabilitation, the study will be explained to his/her proxy and the proxy will receive the informed consent form. Each patient will receive a PIN and all research protocols will be identified only with this PIN. The master list connecting PINs and names will be kept by the rehabilitation facility employee, Dennise Fernandez.
13. The study does not have greater than minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Speaking English

Exclusion Criteria:

* None

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for rehabilitation after a hospitalization
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Rehabilitation time | 30 days
  Actual time spend in rehabilitation
Cooperation with rehabilitation | 30 days
  Willingness to undergo rehabilitation